CLINICAL TRIAL: NCT05691361
Title: A Phase 1, Randomized, Placebo-Controlled, Double-Blind Study in Healthy Volunteers and a Phase 2a, Open-Label Study in Patients With Hereditary Angioedema to Evaluate the Safety, Tolerability, PK and PD of ADX-324
Brief Title: Safety, Tolerability, PK, PD of ADX-324 in Healthy Volunteers and Hereditary Angioedema Patients
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ADARx Pharmaceuticals, Inc. (Industry)
Collaborators: Avance Clinical Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ADX-324-101
Record Dates: First submitted 2022-12-16; First posted 2023-01-20 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Hereditary Angioedema
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — RNA, Small Interfering; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Phase 1, Single-Center, Randomized, Placebo-Controlled, Double Blind Single Ascending Dose Study in HV with expansion into HAE
Who Masked: Participant, Investigator
Masking Description: Double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PART A - Active ADX-324 administered to HV (Experimental): For each cohort in Part A (SAD), 8 participants will be randomized in a 3:1 ratio; 6 participants to active (ADX-324): 2 participants to control (matched placebo). Randomization will be on Day 1. Initially, 2 sentinel participants (1 active and 1 placebo) will be randomized and dosed. The sentinel participants will be evaluated for safety. The investigator's assessment and the independent medical monitor will decide upon the randomization and dosing of the 6 remaining participants (5 active and 1 placebo) according to the randomization schedule.
  Interventions: Drug: ADX-324
- PART A- Placebo administered to HV (Placebo Comparator): For each cohort in Part A (SAD), 8 participants will be randomized in a 3:1 ratio; 6 participants to active (ADX-324): 2 participants to control (matched placebo). Randomization will be on Day 1. Initially, 2 sentinel participants (1 active and 1 placebo) will be randomized and dosed. The sentinel participants will be evaluated for safety. The investigator's assessment and the independent medical monitor will decide upon the randomization and dosing of the 6 remaining participants (5 active and 1 placebo) according to the randomization schedule.
  Interventions: Drug: Placebo
- PART B - ADX-324 administered to HAE participants (Experimental): This will be initiated at the dose level determined by the Safety Review Committee from SAD in HVs. The treatment of HAE participants is an open-label study.
  Interventions: Drug: ADX-324

INTERVENTIONS:
Drug: ADX-324 — siRNA duplex oligonucleotide
  Other Names: siRNA
  Arms: PART A - Active ADX-324 administered to HV; PART B - ADX-324 administered to HAE participants
Drug: Placebo — saline
  Other Names: Saline
  Arms: PART A- Placebo administered to HV

SUMMARY:
The first-in-human Phase 1 study will evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of ADX-324 in healthy volunteers (HV) and in patients with Hereditary Angioedema (HAE).

DETAILED DESCRIPTION:
The clinical study described in this protocol is a Phase 1, single-center study evaluating safety, tolerability, PK, and PD of ADX-324.

The study consists of 2 parts:

* Randomized, double-blind, placebo-controlled, parallel group, single ascending dose (SAD) in HV with up to 6 dose cohorts. For SAD cohorts and planned dosing; and,
* Expansion cohort in participants with Hereditary Angioedema (HAE) at selected dose from Part A and will be open label.

ELIGIBILITY:
Part A - HV

Inclusion Criteria:

1. Male and female adults 18 to 55 years old
2. Body mass index (BMI) between 18 and 30 kg/m2
3. Contraception use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies
4. Willing and able to provide informed consent and comply with all study visits

Exclusion Criteria:

1. Any significant medical history
2. Active malignancy and/or history of malignancy in the past 5 years
3. History of liver disease, Gilbert's syndrome, or abnormal liver function test
4. Estimated creatinine clearance <60 mL/min or serum creatinine > 1.5-fold upper limit of normal.
5. Any active infection or acute illness
6. Major surgery or significant traumatic injury occurring within 3 months
7. Have any other conditions that, in the opinion of the Investigator or Sponsor, would make the participant unsuitable for inclusion, or could interfere with the participant participating in or completing the study.
8. Positive serology tests (HepB, Hep C, HIV)
9. Use of any prescription, vaccines, supplements/vitamins, or over-the counter medication
10. Treatment with another investigational product within 30 days prior to the first study drug administration
11. Known any clinically significant allergic reactions which, in the opinion of the Investigator, would interfere with the volunteer's ability to participate in the study
12. Known hypersensitivity to any of the study drug ingredients.
13. Pregnancy, intent to become pregnant during the course of the study, or lactating women

Part B - HAE

Inclusion Criteria:

1. Male and female ≥18 years old, inclusive, at the time of signing the PICF
2. Confirmed diagnosis of HAE Types I or II
3. Evidence of an average of (at least) one HAE attack per month
4. Participants must have access to, and the ability to use, acute medication(s) to treat angioedema attacks.
5. Body mass index (BMI) between 18 and 30 kg/m2
6. Contraception use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies
7. Willing and able to provide informed consent and comply with all study visits

Exclusion Criteria:

1. Concurrent diagnosis of any other type of chronic angioedema
2. History of clinically significant arterial or venous thrombosis, or current history of a clinically significant prothrombotic risk.
3. Any significant medical history
4. Active malignancy and/or history of malignancy in the past 5 years
5. Any active infection or acute illness, inclusive of cold/flu or COVID-19, within 30 days prior to the first study drug administration.
6. Major surgery or significant traumatic injury occurring within 3 months prior to signature of the PICF
7. Have any other conditions that, in the opinion of the Investigator or Sponsor, would make the participant unsuitable for inclusion, or could interfere with the participant participating in or completing the study.
8. Positive serology tests for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV).
9. Use of C1-INH products, androgens, antifibrinolytics or other small molecule medications for routine prophylaxis within four half-lives prior to screening
10. Must have documented evidence of medical history of HAE attacks
11. Use of any prescription, vaccines, supplements/vitamins, or over-the counter medication (with the exception of oral contraceptives) within 7 days prior to the first study drug administration.
12. Treatment with another investigational product or biologic agent within 30 days prior to the study drug administration
13. History or presence of alcohol abuse or drug use within 30 days prior to the first study drug administration and throughout the study.
14. Blood donation of 50 to 499 mL within 30 days prior to the first study drug administration or of >499 mL within 60 days prior to the first study drug administration.
15. Pregnancy, intent to become pregnant during the course of the study, or lactating women.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Estimated)
Dates: Start 2022-12-14 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety in Healthy Volunteers | 365 days
  To evaluate the safety and tolerability of ADX-324 in HVs by incidence, relationship, and severity of adverse events and serious adverse events
Safety in Healthy Volunteers | 365 days
  To evaluate the safety and tolerability of ADX-324 in HVs by change in baseline electrocardiogram (ECG) parameters (PR, QRS, QT, and QTcF intervals)
Safety in Hereditary Angioedema | 365 days
  To evaluate the safety and tolerability of ADX-324 in HAE by incidence, relationship, and severity of adverse events and serious adverse events

SECONDARY OUTCOMES:
Pharmacokinetics in Healthy Volunteers | 8 days
  To characterize the Pharmacokinetics of ADX-324 in HVs by measuring the Maximum observed concentration (Cmax)
Pharmacokinetics in Healthy Volunteers | 8 days
  To characterize the Pharmacokinetics of ADX-324 in HVs by measuring the Time to Cmax (Tmax)
Pharmacokinetics in Healthy Volunteers | 8 days
  To characterize the Pharmacokinetics of ADX-324 in HVs by measuring the Area under the concentration-time curve from 0 to time of last quantifiable concentration (AUC0-last)
Pharmacokinetics in Healthy Volunteers | 8 days
  To characterize the Pharmacokinetics of ADX-324 in HVs by measuring the Area under the concentration-time curve from 0 to infinity (AUC0-∞)
Pharmacokinetics in Healthy Volunteers | 8 days
  To characterize the Pharmacokinetics of ADX-324 in HVs by measuring the Apparent terminal half-life (t½)
Pharmacokinetics in Healthy Volunteers | 8 days
  To characterize the Pharmacokinetics of ADX-324 in HVs by measuring the Terminal elimination rate constant (λz)
Pharmacokinetics in Healthy Volunteers | 8 days
  To characterize the Pharmacokinetics of ADX-324 in HVs by measuring the Total apparent body clearance (CL/F)
Pharmacokinetics in Healthy Volunteers | 8 days
  To characterize the Pharmacokinetics of ADX-324 in HVs by measuring the Apparent volume of distribution (Vz/F)
Pharmacodynamics in Healthy Volunteers | 365 days
  To characterize the PD of ADX-324 in HVs by the Change from base in plasma concentrations over time of pre Kallikrein (PKK)
Pharmacodynamics in Healthy Volunteers | 365 days
  To characterize the PD of ADX-324 in HVs by the Change from base in plasma concentrations over time of Kallikrein (KK)
Pharmacokinetics in Hereditary Angioedema | 365 days
  To characterize the PD of ADX-324 in HAE by Maximum observed concentration (Cmax) of ADX-324
Pharmacokinetics in Hereditary Angioedema | 8 days
  To characterize the PD of ADX-324 in HAE by Time to Cmax (Tmax) of ADX-324
Pharmacokinetics in Hereditary Angioedema | 8 days
  To characterize the PD of ADX-324 in HAE by Area under the concentration-time curve from 0 to time of last quantifiable concentration (AUC0-last) of ADX-324
Pharmacokinetics in Hereditary Angioedema | 8 days
  To characterize the PD of ADX-324 in HAE by Area under the concentration-time curve from 0 to infinity (AUC0-∞) of ADX-324
Pharmacokinetics in Hereditary Angioedema | 8 days
  To characterize the PD of ADX-324 in HAE by Apparent terminal half-life (t½)
Pharmacokinetics in Hereditary Angioedema | 8 days
  To characterize the PD of ADX-324 in HAE by Terminal elimination rate constant (λz)
Pharmacokinetics in Hereditary Angioedema | 8 days
  To characterize the PD of ADX-324 in HAE by Total apparent body clearance (CL/F)
Pharmacokinetics in Hereditary Angioedema | 8 days
  To characterize the PD of ADX-324 in HAE by Apparent volume of distribution (Vz/F)
Pharmacodynamics in Hereditary Angioedema | 365 days
  To characterize the PD of ADX-324 in HV by Change from base in plasma concentrations over time pre-kallikrein (PKK)
Pharmacodynamics in Hereditary Angioedema | 365 days
  To characterize the PD of ADX-324 in HAE by Change from base in plasma concentrations over time kallikren (KK)

CONTACTS AND LOCATIONS:
Overall Officials: Masako Marai, MD, Study Director — ADARx Pharmaceuticals
Locations (1):
- CMAX Clinical Research, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: Undecided